CLINICAL TRIAL: NCT01575509
Title: A Clinical, Randomized, Comparative Study of Effects of Berry and Grain Products on Postprandial Glycemic Response in Healthy Subjects
Brief Title: A Comparative Study of Effects of Berry and Grain Products on Postprandial Glycemic Response in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Life Sciences Ltd. (Other)
Collaborators: Kiantama Oy (Industry); Suomen Sokeri Oy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MAVI
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Berry product — Sugar infused dried lingonberry
Other: Bread product — Brown bread
Other: Bread product — Whole grain bread
Other: Glucose control solution — Glucose solution with a corresponding amount of carbohydrates as provided by the bread test products
Other: Glucose-fructose control solution — Control solution with a similar carbohydrate content as provided by the dried lingonberry test product

SUMMARY:
This study aims to determine the 2 hour glycemic responses of two bread products and one dried lingonberry product. The average postprandial response of each product is compared with glycemic response after ingestion of control solution with a similar carbohydrate content (glucose, glucose-fructose) as the provided by the respective test product.

ELIGIBILITY:
Inclusion Criteria:

* voluntary given written concent for participation in research
* healthy man or woman, age between 18 and 65 years
* regular eating
* Body Mass Index 18,5 - 29,9 kg/m2

Exclusion Criteria:

* diabetes
* gastrointestinal diseases
* hepatic, kidney, pancreas or thyroid disease or disorder
* arthritis
* pregnancy or breast feeding
* smoking
* allergy
* severe diseases
* blood donation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The 2 hours glycemic responses to test products and control solutions | 2 hours
  Capillary blood samples are taken before and at 15, 30, 45, 60, 90 and 120 min after starting to eat the test products or control solutions for measurements of plasma glucose concentrations.

SECONDARY OUTCOMES:
The 2 hours insulinemic responses to dried lingonberry product and corresponding control solution | 2 hours
  Capillary blood samples are collected before and at 15, 30, 45, 60, 90 and 120 min after eating the lingonberry test product and glucose-fructose control solution. The serum insulin concentrations are analysed.
The incremental area under glucose curve (IAUC) of bread test products | 2 hours
  IAUC (mmol/l x min) is determined using the trapezoidal method for each subject and bread test product and corresponding glucose control solution.
Glycemic index (GI) of bread test products
  The GI is calculated as a percentage of the glucose IAUC values of a bread product and a glucose control solution.

CONTACTS AND LOCATIONS:
Overall Officials: Päivi Cheney, MD, Principal Investigator
Locations (1):
- Clinical Life Sciences Ltd, Kajaani, Finland